CLINICAL TRIAL: NCT03329027
Title: A Prospective, Multicenter, Randomized, Double-blind, Sham-controlled Pilot Study to Assess the Efficacy and Safety of Various Vibrating Capsule Modes
Brief Title: A Pilot Study to Assess the Efficacy and Safety of Various Vibrating Capsule Modes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300CLD
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active Comparator-Vibrating Mode 1 (Experimental): Patients will receive vibrating capsule Vibrating Mode 1 for 8 weeks of treatment (5 capsules/week). Active Mode 1 and Active Mode 2 differ in their vibration sessions
  Interventions: Device: Vibrating Capsule
- Active Comparator-Vibrating Mode 2 (Experimental): Patients will receive vibrating capsule Vibrating Mode 2 for 8 weeks of treatment (5 capsules/week). Active Mode 1 and Active Mode 2 differ in their vibration sessions
  Interventions: Device: Vibrating Capsule
- Sham Comparator (Sham Comparator): Patients will receive sham capsule for 8 weeks of treatment (5 capsules/week). The Sham capsule is visually similar to the active capsules (Active Mode 1 and Active Mode 2, which differ in their vibration sessions) but without the active components.
  Interventions: Device: Sham capsule

INTERVENTIONS:
Device: Vibrating Capsule — Patients will receive vibrating capsule for 8 weeks of treatment (5 capsules/week)
  Arms: Active Comparator-Vibrating Mode 1; Active Comparator-Vibrating Mode 2
Device: Sham capsule — Patients will receive vibrating capsule for 8 weeks of treatment (5 capsules/week)
  Arms: Sham Comparator

SUMMARY:
The study is a prospective, adaptive, multicenter, randomized, double-blind, Sham-controlled pilot study, to evaluate the efficacy and safety of the Vibrant Capsule in relieving constipation in subjects with functional constipation.

Three arms that assessed:

* Vibrant Capsule with vibrating mode 1 administered 5 times per week
* Vibrant Capsule with vibrating mode 2 administered 5 times per week
* Sham Capsule administered 5 times per week

DETAILED DESCRIPTION:
Subjects will be followed continuously for at least a 2 weeks run-in period and then be randomized to either Vibrant or Sham capsules for a treatment period of 8 weeks. The first 2 weeks of treatment will be considered as a subjects' training period.

Data reporting will be done on an electronic Case Report Form and an eDiary. Subjects will be asked to refrain from taking any medication or supplement to relieve their constipation, during the entire study period.

After the run-in period, the subjects will return and eligibility will be re-assessed. Subjects will be trained on how to use the base unit and will swallow the first capsule on site the day of baseline visit. They will activate and ingest the rest of the capsules at home by themselves, using the base unit.

Subjects will be instructed to complete a simple subject eDiary each day throughout the duration of the study. A final visit will take place at the end of the 8 week treatment period.

Subjects will receive phone calls at least once a week and subject compliance will be monitored during the 8 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 22 years and older
* Subjects with Chronic Idiopathic Constipation according to Rome III criteria and who have not experienced relief of their symptoms from available therapies
* Subjects with an average of <3 Spontaneous Bowel Movements per week and ≥1 Spontaneous Bowel Movements per week
* Normal colonoscopy performed within 10 years prior to study participation, unless the subjects are <50 years old and without alarm signs and/or symptoms
* Subject signed the Informed Consent Form
* Female subjects must have a negative pregnancy test

Exclusion Criteria:

* History of complicated/obstructive diverticular disease
* History of intestinal or colonic obstruction, or suspected intestinal obstruction.
* History of significant gastrointestinal disorder, including any form of inflammatory bowel disease or gastrointestinal malignancy
* History of gastroparesis
* Use of any of the following medications:
* Medications that may affect intestinal motility, prokinetics, anti-Parkinsonian medications, opiates, opioids, calcium-channel blockers, aluminum/magnesium hydroxide
* With the exception of antidepressants, thyroid or hormonal replacement therapy, when the subject has been on a stable dose for at least 3 months prior to enrollment.
* Clinical evidence of significant respiratory, cardiovascular, renal, hepatic, biliary, endocrine, psychiatric or neurologic disease.
* Presence of cardiac pacemaker or gastric electrical stimulator.
* History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
* Diagnosis of mega-rectum or colon, congenital anorectal malformation, clinically significant rectocele, history of intestinal resection (with an exception for appendectomy, cholecystectomy and inguinal hernia repair), history of bariatric surgery or evidence of any structural abnormality of the gastrointestinal tract that might affect transit
* History of Zenker's diverticulum, dysphagia, Barrett's esophagus, esophageal stricture or achalasia
* Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Subjects with pelvic floor dysfunction/defecatory disorder
* Participation in another clinical study within one month prior to screening.
* Women who are pregnant or lactating

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Malina, B.SC MBA, Study Director — Vibrant Gastro
Locations (4):
- United States (4):
  - Hope Clinical Research, Canoga Park, California
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Great Lakes Medical Research, Willoughby, Ohio
  - Health Research of Hampton Roads, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No
Data from this study will be presented in future Vibrantgastro publications.

RESULTS

PARTICIPANT FLOW:
Groups:
- Vibrant Active Mode 1; Vibrant Active Mode 2: Patients will receive vibrating capsule for 8 weeks of treatment (5 capsules/week)
  Vibrating Capsule: Patients will receive vibrating capsule for 8 weeks of treatment (5 capsules/week)
- Sham: Patients will receive sham capsule for 8 weeks of treatment (5 capsules/week)
  Sham capsule: Patients will receive vibrating capsule for 8 weeks of treatment (5 capsules/week)
Period: Overall Study
Arm/Group | Vibrant Active Mode 1 | Vibrant Active Mode 2 | Sham
Started | 21 | 22 | 24
Completed | 11 | 17 | 16
Not Completed | 10 | 5 | 8
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 9 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibrant Active Mode 1 | Vibrant Active Mode 2 | Sham | Total
Number analyzed (Participants) | 21 | 22 | 24 | 67
Age, Customized [Mean (Full Range); unit: years]
  Age | 44.39 [25.56 to 68.00] | 41.85 [24.31 to 60.25] | 41.31 [22.05 to 66.59] | 42.51 [22.05 to 68.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 21 | 57
  Male | 3 | 4 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 5 | 9 | 20
  Hispanic or Latino | 4 | 8 | 6 | 18
  Black or African American | 10 | 7 | 9 | 26
  Native American or American Indian | 1 | 1 | 0 | 2
  Asian/ Pacific Islander | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 22 | 24 | 67
Duration of constipation [Mean (Full Range); unit: years] | 14.86 [2 to 47] | 8.45 [1 to 30] | 11.15 [0.5 to 52] | 11.48 [0.5 to 52]

OUTCOME MEASURES:

1. Primary Outcome: CSBM1- an Increase of at Least One Weekly Complete Spontaneous Bowel Movement (CSBM) During at Least 6 of the 8 Weeks of Treatment
Description: CSBM1 success rate, defined as an increase from the base line of at least one weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment
Time Frame: 8 weeks
Population: Analysis of 44 subjects who completed at least 6 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator-Vibrating Mode 1 | Active Comparator-Vibrating Mode 2 | Sham Comparator
Number analyzed (Participants) | 11 | 17 | 16
Participants | 7 | 7 | 9

2. Primary Outcome: CSBM2- an Increase of at Least Two Weekly Complete Spontaneous Bowel Movement (CSBM) During at Least 6 of the 8 Weeks of Treatment
Description: CSBM2 success rate, defined as an increase from the base line of at least two weekly Complete Spontaneous Bowel Movement (CSBM) during at least 6 of the 8 weeks of treatment.
Time Frame: 6-8 weeks
Population: Analysis of 44 subjects who completed at least 6 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Active Mode 1 | Vibrant Active Mode 2 | Sham
Number analyzed (Participants) | 11 | 17 | 16
Participants | 2 | 4 | 6

3. Secondary Outcome: SBM 1- Success Rate, Defined as as an Increase From the Base Line of at Least One Weekly Spontaneous Bowel Movement (SBM) During at Least 6 of the 8 Weeks of Treatment.
Description: SBM success rate, defined as as an increase from the base line of at least one weekly Spontaneous Bowel Movement (SBM) during at least 6 of the 8 weeks of treatment. Subjects with less than 2 weeks (with at least 5 days per week) of valid diary during the treatment period will be considered as non-evaluable.
Time Frame: 6-8 weeks
Population: Analysis of 44 subjects who completed at least 6 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrant Active Mode 1 | Vibrant Active Mode 2 | Sham
Number analyzed (Participants) | 11 | 17 | 16
Participants | 8 | 9 | 7

ADVERSE EVENTS:
Time Frame: For each patient, safety data was collected for 10 weeks of study participation.
Arm/Group | Vibrant Active Mode 1 | Vibrant Active Mode 2 | Sham
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 4/21 | 7/22 | 5/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vibrant Active Mode 1 (N=21) | Vibrant Active Mode 2 (N=22) | Sham (N=24)
Abdominal pain/discomfort (Gastrointestinal disorders) | 1 | 2 | 0 — Abdominal pain/discomfort
Abdominal distention/Bloating and/or Flatulence (Gastrointestinal disorders) | 2 | 1 | 0 — Abdominal distention/Bloating and/or Flatulence
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 — Diarrhea
Sensation of vibration (Product Issues) | 1 | 2 | 3 — Sensation of vibration
UTI (Renal and urinary disorders) | 0 | 1 | 0 — Urinary Tract Infection\Cystitis
Headache (General disorders) | 1 | 3 | 1 — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT03329027/Prot_SAP_000.pdf